CLINICAL TRIAL: NCT06580652
Title: Measurement of Tidal Volumes Achieved With Tracheal Tubes and Laryngeal Mask Airways During in Hospital Cardiac Arrest.
Brief Title: Respiratory Parameters Using Advanced Airways During In-hospital Cardiac Arrest
Status: Recruiting | Type: Observational
Sponsor: Royal United Hospitals Bath NHS Foundation Trust (Other)
Collaborators: RCUK (Unknown)
Responsible Party: Sponsor
Other Study IDs: 328233
Record Dates: First submitted 2024-03-12; First posted 2024-08-30 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tracheal Tube: participants in cardiac arrest in whom a tracheal tube is used as the airway device
- Supraglottic Airway: participants in cardiac arrest in whom a supraglottic airway is used as the airway device

SUMMARY:
The investigators aim to investigate the real life volumes of air delivered to the lungs when rescuers deliver these breaths by hand as part of resuscitation attempts during cardiac arrest. The study will compare the volumes achieved using different devices which are routinely used to provided an airway during routine cardiac arrest care. Volumes will be measured using a small non intrusive device which sits in the airway circuit and measures flow of air in real time. The patients chosen for this study will be those already recruited to an ongoing trial (AIRWAYS-3) assessing the outcomes for patients suffering in hospital cardiac arrest based on airway device used.

DETAILED DESCRIPTION:
Patients meeting the AIRWAYS-3 inclusion criteria will be enrolled. Aged > 18, undergoing cardiopulmonary resuscitation and a clinician present able to perform both tracheal intubation and insertion of an SGA.

Patients in the emergency department, patients under 18 and pregnant patients will excluded. Patients will be treated exactly as per the AIRWAYS-3 protocol.

Following randomisation a VFD device will be placed in the breathing system (Figure 2). The device will be left in situ until manual ventilation ceases during the IHCA event. The VFD will be used with the screen deactivated so as not to affect the airways rescuers normal practice. Cessation of manual ventilation may occur for the following reasons: patient resumed breathing spontaneously, use of mechanical ventilator, decision to stop resuscitation event (death).

Anonymised ventilation data will be downloaded following each IHCA event. The following data will be collected alongside from the existing NCAA data and AIRWAYS-3 CRF.

* Age
* Actual Weight (kg) - Measured or estimated
* Height (cm)
* Gender (M/F)
* Calculated Ideal Body Weight (kg)
* Duration of arrest
* Presenting rhythm
* Outcome of arrest - dead/alive
* Recorded respiratory disease
* Timeline of airway insertion events
* Advanced airway arm

Respiratory data to be collected from VFD:

* Duration of intervention
* Average TV (ml)
* Largest TV (ml)
* Smallest TV (ml)
* Average (mean) leak volume (ml)
* Average respiratory rate
* Average (mean) inspiratory time (s)
* Average (mean) expiratory time (s)

Mean and range values will be recorded for each parameter and grouped according to advanced airway device used.

Data will be analysed using a commercial statistical software package. Descriptive and comparative statistical calculations will be performed including mean/median average, standard deviation, correlation, the Chi Square and Student t tests. Correlations and predictions will include regression analysis, Wilcoxon Rank Sum and ANOVA. If more advanced statistical analysis is required (the need for which will be based on the results from the simple statistical calculations and quality of data obtained), then a formal statistical consult will be sought from the Warwick Clinical Trials Unit.

Sample Size A power calculation has been completed. Experimental bench data suggests manual bag ventilation achieved tidal volumes of 480ml during cardiopulmonary resuscitation. Based on a mean tidal volume of 500ml to detect a minimal difference of 100ml with a standard deviation of 100ml with power set at 80% and significance of 0.05. The study will require 15 participants per group. Total sample size = 30.

ELIGIBILITY:
Inclusion Criteria:

* As per AIRWAYS-3 trial:
* In-hospital cardiac arrest, attended by the hospital cardiac arrest team in response to a cardiac arrest call (2222 or equivalent), and when a clinician permitted to undertake both tracheal intubation and supraglottic airway placement (so that either intervention can be delivered) is present
* Undergoing resuscitation and requiring advanced airway management in the opinion of the trained clinician responsible for randomisation

Exclusion Criteria:

* As per AIRWAYS-3 trial
* Patients who have a cardiac arrest outside hospital and who are transported to the hospital in ongoing cardiac arrest
* People who are not a hospital inpatient (e.g. visitor, relative, staff or outpatient)
* Patients who are already tracheally intubated at the time of eligibility assessment
* Patients known to be pregnant
* Patients with a functioning tracheostomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered a cardiac arrest whilst an in patient.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Tidal Volume | assessed from the initiation of advanced airway management to the cessation of the resuscitation treatment (Return of spontaneous circulation or death). Through completion of data collection, ranging between minutes to 1 hour.
  The mean tidal volume achieved during cardiac arrest treatment

SECONDARY OUTCOMES:
Mean leak | assessed from the initiation of advanced airway management to the cessation of the resuscitation treatment (Return of spontaneous circulation or death). Through completion of data collection, ranging between minutes to 1 hour.
  The mean volume of leak recorded during cardiac arrest treatment
inspiratory time | assessed from the initiation of advanced airway management to the cessation of the resuscitation treatment (Return of spontaneous circulation or death). Through completion of data collection, ranging between minutes to 1 hour.
  The mean inspiratory time during cardiac arrest treatment
Expiratory time | assessed from the initiation of advanced airway management to the cessation of the resuscitation treatment (Return of spontaneous circulation or death). Through completion of data collection, ranging between minutes to 1 hour.
  The mean expiratory time during cardiac arrest treatment

OTHER OUTCOMES:
Respiratory rate | assessed from the initiation of advanced airway management to the cessation of the resuscitation treatment (Return of spontaneous circulation or death). Through completion of data collection, ranging between minutes to 1 hour.
  Mean Respiratory rate delivered during cardiac arrest treatment
Smallest tidal volume | assessed from the initiation of advanced airway management to the cessation of the resuscitation treatment (Return of spontaneous circulation or death). Through completion of data collection, ranging between minutes to 1 hour.
  The smallest tidal volume delivered during cardiac arrest treatment
largest tidal volume | assessed from the initiation of advanced airway management to the cessation of the resuscitation treatment (Return of spontaneous circulation or death). Through completion of data collection, ranging between minutes to 1 hour.
  The largest tidal volume delivered during cardiac arrest treatment
duration of intervention | assessed from the initiation of advanced airway management to the cessation of the resuscitation treatment (Return of spontaneous circulation or death). Through completion of data collection, ranging between minutes to 1 hour.
  The time for which the airway device was used during cardiac arrest treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Spencer, Study Chair — Royal United Hosptial Bath
Locations (1):
- Royal United Hospital Bath, Bath, Banes, United Kingdom

IPD SHARING:
Plan to Share IPD: No